CLINICAL TRIAL: NCT02159443
Title: Characterization of Pretreatment Anti-Therapeutic Antibodies (PATA) in Patients Treated With hu14.18K322A Antibody
Brief Title: Pretreatment Anti-Therapeutic Antibodies (PATA) in Patients Treated With hu14.18K322A Antibody
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: PATA
Record Dates: First submitted 2014-06-05; First posted 2014-06-10 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Ewing Family of Tumors; Melanoma; Neuroblastoma; Osteosarcoma
Keywords: Hu14.18K322A; Human anti-human antibodies (HAHA); Pretreatment anti-therapeutic antibodies (PATA)
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive, Peripheral; Melanoma; Neuroblastoma; Osteosarcoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from tumor tissue. Blood serum samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Participants: Those who meet eligibility criteria and consent to participate in the study.

SUMMARY:
Hu14.18K322A is a monoclonal antibody developed at St. Jude Children's Research Hospital (SJCRH) that is made to bind to cancer cells that have a molecule called GD2 on their surface. Sometimes the human body will make an antibody to the therapeutic antibody (like hu14.18K322A) that is being given for treatment. These are called human anti-human antibodies (HAHA). When testing for HAHA in a previous cohort of patients who received hu14.18K322A, it was found that some patients tested positive for high levels of an antibody before receiving hu14.18K322A or any other anti-GD2 antibody. In this study, investigators would like to know more about the nature of this pretreatment antibody, how often is it present, and if in the laboratory it increases the killing of tumor cells.

OBJECTIVES:

* To determine whether pretreatment anti-therapeutic antibodies (PATA) represent antibodies reactive against an epitope (allotypic determinant) found on the anti-GD2 antibody hu14.18K322A
* To determine if PATA increases the anti-tumor efficacy of anti-GD2 antibodies in vitro

DETAILED DESCRIPTION:
In the proposed study, investigators will seek to determine the nature of this antibody that is being detected in the HAHA test for this group of patients, and if, in the laboratory, it increases the killing of tumor cells, accounting for the observation that some the patients who tested positive may have an improved outcome.

The study will analyze DNA from blood samples of SJCRH patients treated with hu14.18K322A anti-GD2 antibody. Serological studies and confirmatory genotyping studies will be performed in a laboratory at the University of Wisconsin.

ELIGIBILITY:
Inclusion Criteria:

* All participants who have or will receive treatment at SJCRH with hu14.18K322A.

Exclusion Criteria:

* Those not receiving treatment at SJCRH with hu14.18K322A.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will have a diagnosis within the Ewing family of tumors, melanoma, neuroblastoma, or osteosarcoma and will receive treatment with hu14.18K322A.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2014-07-15 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2020-04-24 (Actual)

PRIMARY OUTCOMES:
Characterization of PATA | Once at participant enrollment
  Objective: To determine whether pretreatment anti-therapeutic antibodies (PATA) represent antibodies reactive against an epitope (allotypic determinant) found on the anti-GD2 antibody hu14.18K322A
Number of samples with increased anti-tumor efficacy | Once, at enrollment
  Objective: To determine if PATA increases the anti-tumor efficacy of anti-GD2 antibodies in vitro

CONTACTS AND LOCATIONS:
Overall Officials: Victor Santana, MD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude Children's Research Hospital — http://www.stjude.org/protocols